CLINICAL TRIAL: NCT05275569
Title: Personalized Electroacupuncture Treatment Combined With Standard Antiemetic Drugs for Chemotherapy-induced Nausea and Vomiting in Patients With Breast Cancer Receiving Highly Emetogenic Chemotherapy
Brief Title: Personalized Electroacupuncture Treatment for Chemotherapy-induced Nausea and Vomiting in Breast Cancer (PET)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHQU-2022002
Record Dates: First submitted 2022-01-25; First posted 2022-03-11 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: electroacupuncture treatment; chemotherapy-induced nausea; chemotherapy-induced vomiting; breast cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True acupuncture + standard antiemetic treatment (Experimental)
  Interventions: Procedure: True acupuncture + standard antiemetic treatment
- Sham acupuncture + standard antiemetic treatment (Placebo Comparator)
  Interventions: Procedure: Sham acupuncture + standard antiemetic treatment

INTERVENTIONS:
Procedure: True acupuncture + standard antiemetic treatment — Participants will receive electroacupuncture once daily from day 1 to day 4. The acupuncturists will insert needles into the acupoints and manipulate the needles until"de qi"sensation is achieved and reported by the participants. Electrical stimulation will be delivered for 30 minutes at alternating frequencies of 2/10Hz. They will receive fosaprepitant 150 mg intravenous IV + palonosetron 0.25 mg IV + dexamethasone 10 mg IV 30 minutes prior to chemotherapy on Day 1, dexamethasone 8 mg IV on days 2, 3, 4 post chemotherapy.
  Arms: True acupuncture + standard antiemetic treatment
Procedure: Sham acupuncture + standard antiemetic treatment — The sham acupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive minimal acupuncture treatment without electrical stimulation at the same time as the intervention group.Care was taken to avoid "de qi" sensation. They will receive fosaprepitant 150 mg intravenous IV + palonosetron 0.25 mg IV + dexamethasone 10 mg IV 30 minutes prior to chemotherapy on Day 1, dexamethasone 8 mg IV on days 2, 3, 4 post-chemotherapy(the antiemetic drugs are the same as the true acupuncture group).
  Arms: Sham acupuncture + standard antiemetic treatment

SUMMARY:
This study aims to evaluate electroacupuncture as an antiemetic treatment compared with sham acupuncture in patients with breast cancer, receiving highly emetogenic chemotherapy (HEC). Moreover, it will analyze the association between single nucleotide polymorphism and the antiemetic outcomes of electroacupuncture.

DETAILED DESCRIPTION:
This is a parallel-group, triple-blinded (participants, evaluators and statisticians), randomized controlled study that investigates the antiemetic role of electroacupuncture combined with standard antiemetic drugs for patients with breast cancer receiving HEC. Neurokinin-1 receptor antagonists (NK-1RAs), serotonin receptor antagonists [5HT3RA] and dexamethasone will be administered prior to initiation of HEC on Day 1 in both groups. Electroacupuncture or sham acupuncture will be randomly administered to the two groups. Subjects will record all events of emesis and the use of rescue antiemetic medication for nausea and/or vomiting. Blood samples will be collected and be analyzed to whether genetic polymorphisms can be used to predict Electroacupuncture outcomes in patients with breast cancer receiving HEC. Primary and secondary outcomes and adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, of any nationality;
2. Eastern Cooperative Oncology Group performance status of 0-2;
3. For patients with breast cancer, molecular typing is not limited, receiving for the first time chemotherapy with anthracyclines+ cyclophosphamide (EC or AC) or carboplatin (AUC≥4)/cisplatin -based HEC regimen. Patients with previous chemotherapy use could be enrolled if they received it >3 months;
4. Predicted life expectancy of ≥3 months;
5. Adequate bone marrow, kidney, and liver function;
6. Adequate contraception if premenopausal women;
7. Written informed consent by the patient before enrolment.

Exclusion Criteria:

1. Patients already submitted to chemotherapy;
2. Is scheduled to receive any non-HEC on Day 1;
3. Received or is scheduled to receive radiation therapy to the abdomen, pelvis, head and neck within 1 week prior to Day 1 or between Days 1 to 5 in cycle 1;
4. Has symptomatic primary or metastatic symptomatic central nervous system malignancy causing nausea and/or vomiting;
5. Have ongoing emesis or CTCAE grade 2 or greater nausea;
6. Significant mental conditions;
7. Any allergies to study drug, antiemetics or dexamethasone;
8. Significantly abnormal laboratory values (platelets, absolute neutrophils, AST, ALT, bilirubin or creatinine);
9. Patients who are pregnant or breast-feeding;
10. Inflammatory skin reaction;
11. Has lymphedema in acupuncture stimulation area;
12. Patients who are afraid of electroacupuncture stimulation or allergic to stainless steel needles;
13. Received acupuncture treatments for any conditions less than 4 weeks before HEC;
14. The current use of any drugs with antiemetic activity (e.g. 5-HT3 RA, dopamine receptor antagonist, minor tranquilizer, antihistamine);
15. Patients with concomitant severe diseases or with a predisposition to emesis such as gastrointestinal obstruction, active peptic ulcer, hypercalcemia and symptomatic brain metastasis;
16. Patients receiving other concomitant antiemetic treatments or submitted to antiemetic treatments in the 24 hours before chemotherapy;
17. Patients receiving concomitant steroids, except when administered at physiologic doses;
18. Patients receiving concomitant benzodiazepines, except when used for nocturnal sedation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients With Significant Nausea, Rescue Treatment and Number of Times of Vomiting Occurs After chemotherapy (complete protection). | 120 hours
  The proportion of patients achieving complete protection is defined as patients who have no vomiting, no rescue treatment, no significant nausea that was assessed by visual analog scale (VAS, this is a Visual Analogue Scale was used to assess the incidence and intensity of nausea daily, a 100-mm horizontal bar containing no marking except for the anchor point at each end: left, no nausea; right, worst nausea. No nausea was defined as a VAS scores < 5mm, no significant nausea was defined as a VAS scores < 25mm), and maximum less than 25 mm during the first 120 hours after the initiation of chemotherapy (The definition is different from the complete response in the "Secondary endpoints" section).

SECONDARY OUTCOMES:
The relationship between single nucleotide polymorphism genotypes and the proportion of patients with significant nausea, rescue treatment and number of times of vomiting occurs after chemotherapy (complete protection). | 120 hours
  The single nucleotide polymorphism genotypes will be analyzed by detecting different bases (A, T, C and G) in peripheral blood DNA. The proportion of patients with different single nucleotide polymorphism genotypes will be analyzed. The proportion of patients achieving complete protection is defined as patients who have no vomiting, no rescue treatment, no significant nausea that was assessed by VAS as mentioned above, and maximum less than 25 mm during the first 120 hours after the initiation of chemotherapy. We will analyze the relationship between the proportion of patients with different single nucleotide polymorphism genotypes and the proportion of patients with complete protection.
The proportion of patients who have no vomiting/retching or rescue medications after chemotherapy during 0 to 24 hours (acute complete response) | 24 hours
  The proportion of patients achieving acute complete response is defined as patients who have no vomiting/retching or rescue medications during 0 to 24 hours after the initiation of chemotherapy.
The proportion of patients who have no vomiting/retching or rescue medications after chemotherapy during 24 to 120 hours (delayed complete response) | 120 hours
  The proportion of patients achieving delayed complete response is defined as patients who have no vomiting/retching or rescue medications during delayed 24 to 120 hours after the initiation of chemotherapy.
Number of times of no vomiting in the acute stage (0 to 24 hours) after chemotherapy (no vomiting in the acute stage) | 24 hours
  The proportion of patients who have no vomiting during the acute stage (0 to 24 hours) after the initiation of chemotherapy.
Number of times of no vomiting in the delayed stage (24 to 120 hours) after chemotherapy (no vomiting in the delayed stage) | 120 hours
  The proportion of patients who have no vomiting during the delayed stage (24 to 120 hours) after the initiation of chemotherapy.
Number of times of no vomiting in the overall stage (0 to 120 hours) after chemotherapy (no vomiting in the overall stage) | 120 hours
  The proportion of patients who have no vomiting during 0 to 120 hours after the initiation of chemotherapy.
The proportion of no nausea (no nausea in the overall stage) | 120 hours
  The proportion of patients who have no nausea (VAS# 5 mm) that was assessed by VAS, and maximum less than 5 mm during the first 120 hours after the initiation of chemotherapy.
The proportion of no significant nausea (no significant nausea in the overall stage) | 120 hours
  The proportion of patients who have no significant nausea (VAS# 25 mm) that was assessed by VAS, and maximum less than 25 mm during the first 120 hours after the initiation of chemotherapy.
The proportion of patients achieving total control (total control in the overall stage) | 120 hours
  The proportion of patients achieving total control is defined as patients who have no vomiting, no rescue treatment, no nausea assessed by VAS, and maximum less than 5 mm during the first 120 hours after the initiation of chemotherapy.
Constipation | 120 hours
  The proportion of patients with constipation evaluated by Common Terminology Criteria for adverse events Version 4.0 during 0 to120 hours after the initiation of chemotherapy.
Diarrhea | 120 hours
  The proportion of patients with diarrhea evaluated by Common Terminology Criteria for adverse events Version 4.0 during 0 to120 hours after the initiation of chemotherapy.
Fatigue | 120 hours
  The proportion of patients with fatigue evaluated by Common Terminology Criteria for adverse events Version 4.0 during 0 to120 hours after the initiation of chemotherapy.
Insomnia | 120 hours
  The proportion of patients with insomnia evaluated by Common Terminology Criteria for adverse events Version 4.0 during 0 to120 hours after the initiation of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiuda Zhao, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen G, Ren D, Zhao F, Wang M, Liu Z, Feng X, He Y, Liu X, Ling X, Zhao Y, Song F, Ma J, Li E, She T, Liu Z, Li Z, Huang S, Chen Y, Yang J, Li X, Duan L, Da M, Zheng Y, Li Y, Zhao J. Effect of Adding Electroacupuncture to Standard Triple Antiemetic Therapy on Chemotherapy-Induced Nausea and Vomiting: A Randomized Controlled Clinical Trial. J Clin Oncol. 2024 Dec;42(34):4051-4059. doi: 10.1200/JCO.24.00099. Epub 2024 Sep 6. PMID 39241208